CLINICAL TRIAL: NCT06425718
Title: Comparison of Transversalis Fascia Plane Block and Surgical Site Local Anesthetic Infiltration in Elective Cesarean Section Surgeries
Brief Title: Comparison of Postoperative Analgesia Methods in Elective Cesarean Section Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: MarmaraClinical
Record Dates: First submitted 2024-04-26; First posted 2024-05-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Opioid Use; Postoperative Pain
Keywords: opioid use; postoperative pain; transversalis plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversalis Fascia Plane Block (Active Comparator): Bilateral Transversalis Fascia Plane Block (with %0.25 bupivacaine, 20 ml for each side) and intravenous tramadol via Patient Controlled Analgesia device (5 mg/ml tramadol, bolus dose: 1ml, lock time: 10 minutes)
  Interventions: Procedure: Postoperative Pain Management Technique
- Surgical Site Local Anesthetic Infiltration (Active Comparator): Local anesthetic infiltration will be applied to the surgical incision area with 0.25% 20 ml bupivacaine and intravenous tramadol via Patient Controlled Analgesia device (5 mg/ml tramadol, bolus dose: 1ml, lock time: 10 minutes)
  Interventions: Procedure: Postoperative Pain Management Technique

INTERVENTIONS:
Procedure: Postoperative Pain Management Technique — Patients who will undergo cesarean section under spinal anesthesia will be included. Comparing postoperative pain and opioid consumption in groups

SUMMARY:
Since many intravenous anesthetic agents administered to the mother can cross the placental barrier and cause fetal side effects, multimodal analgesia strategies with peripheral nerve blocks are preffered with greater safety in elective Cesarean section surgeries.

The primary objective of this study is to compare postoperative opioid consumption and pain scores (NRS) in elective cesarean section patients who receive a transversalis fascia plane block versus those who receive surgical site local anesthetic infiltration in addition to spinal anesthesia.

DETAILED DESCRIPTION:
After Cesarean sections, several factors play a role in the formation of postoperative pain, including parietal stimulation originating from the surgical incision, visceral stimulation originating from the peritoneum, and manipulation of intra-abdominal structures.

To enhance patients' rehabilitation during the postoperative period, promote lactation and infant care, and reduce hospital stays, the most appropriate postoperative analgesia method should be selected.

Since many intravenous anesthetic agents administered to the mother can cross the placental barrier and cause fetal side effects, regional anesthesia techniques are preferred with greater safety in elective Cesarean section surgeries.

In the postoperative period, multimodal analgesia strategies can be used for pain control, and one of these strategies is postoperative peripheral nerve blocks. Ultrasound guided transversalis fascia plane block is one of the preferred methods for postoperative analgesia in cesarean section patients.

The primary objective of this study is to compare postoperative opioid consumption and pain scores (NRS) in elective cesarean section patients who receive a transversalis plane block versus those who receive surgical site local anesthetic infiltration in addition to spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* ASA II-III patients undergoing elective cesarean section

Exclusion Criteria:

* ASA IV patients
* Patients with known neurologic or psychiatric disorders
* Patients with clinically significant cardiovascular, respiratory, hepatic, renal or metabolic disease
* Patients with alcohol or drug addiction
* Mentally disabled patients
* Patients with BMI>30
* Patients who develop massive bleeding or coagulopathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Comparison of postoperative opioid consumption between two groups via Patient Controlled Analgesia (PCA) device | 24 hours
  Intravenous patient-controlled analgesia (PCA) is a system of opioid delivery that consists of an infusion pump interfaced with a timing device. Intravenous tramadol consumption will be recorded via PCA device, then it will be documented in mg/kg units.

SECONDARY OUTCOMES:
Postoperative pain assessment with Numeric Rating Scale (NRS) | 24 hours
  In a Numerical Rating Scale (NRS), patients are asked to choose from 1 to 10. 1: no pain 10: worst pain experienced

CONTACTS AND LOCATIONS:
Overall Officials: Beliz Bilgili, Principal Investigator — Marmara University
Locations (1):
- Marmara University Pendik Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided